CLINICAL TRIAL: NCT06860412
Title: Efficacy of a Dog Assisted Group Intervention in Elderly People with Unwanted Loneliness: Project "Paws with You"
Brief Title: Efficacy of a Dog Assisted Group Intervention in Elderly with Unwanted Loneliness
Acronym: AAI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Loneliness 25/020-P
Record Dates: First submitted 2025-03-04; First posted 2025-03-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Loneliness; Elderly (people Aged 65 or More); Animal Assisted Therapy
Keywords: Animal Assisted Therapy; Elderly; Loneliness; Social isolation; Primary Healthcare; Human-Animal Interactions
MeSH Terms: conditions — Social Isolation; Human-Animal Interaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The principal statistician are blind to identifying participant information and group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Animal Assisted Intervention (Experimental): Participants assigned to the experimental arm will receive active non-pharmacological treatment utilizing a Psychoeducational Intervention accompanied by live therapy dogs. The experimental group will carry out a total of 9 group sessions of one and a half hour duration, on a weekly basis for 9 consecutive weeks. The groups will be formed by 10 participants.
  Interventions: Behavioral: Animal Assisted Intervention
- Psychoeducational Intervention as Usual (Active Comparator): Participants assigned to the active comparator arm will receive active non-pharmacological treatment utilizing a psychoeducational intervention as usual. The participants carry out a total of 9 group sessions of one and a half hour duration, on a weekly basis for 9 consecutive weeks. The groups will be formed by 10 participants.
  Interventions: Behavioral: Psychoeducational Intervention as Usual

INTERVENTIONS:
Behavioral: Animal Assisted Intervention — This is a multimodal group intervention program that simultaneously carries out health education activities, physical activities, emotional activities and social interactions through the integration of a psychoeducational intervention and animal-assisted therapy for elderly people with unwanted loneliness.
  Arms: Animal Assisted Intervention
Behavioral: Psychoeducational Intervention as Usual — This psychoeducational intervention is a multimodal group intervention program that simultaneously carries out health education activities, physical activities, emotional activities and social interactions for elderly people with unwanted loneliness.
  Arms: Psychoeducational Intervention as Usual

SUMMARY:
The purpose of this study is to evaluate the efficacy of a dog-assisted group intervention in elderly people with unwanted loneliness; in terms of improving the perception of unwanted loneliness and emotional well-being. To analyze whether differences are obtained in social support and to determine the satisfaction of the participants. Participants will be recruited from a Primary Health Care Center. These objectives will be accomplished through a randomized clinical trial, single blind, two-arm study of AAT for elderly people with unwanted loneliness.

DETAILED DESCRIPTION:
Background: Unwanted loneliness negatively affects the physical and psychological health of older adults, as well as increasing the likelihood of engaging in behaviors harmful to health. This is an increasing reality and is considered a public health problem. Animal-Assisted Therapy (AAT) is a planned, structured, goal-oriented therapeutic intervention directed by health professionals.

Purposes: To evaluate the efficacy of AAT (with therapy dogs) in elderly people with unwanted loneliness. To assess whether there are differences in the scores obtained after the group intervention regarding the perception of unwanted loneliness and emotional well-being. To analyze whether differences are obtained in social support. To determine participants' satisfaction with the group intervention.

Methodology: A two-arm randomized controlled clinical trial (control group (CG) and experimental group (EG)) with a simple blind (evaluator). Participants will be recruited from a Primary Health Care Center: aged 65 or older, diagnosed as "living alone," and experiencing unwanted loneliness. Intervention: The EG will participate in 9 psycho-educational group sessions (once-a week, 90 minutes) with a therapy dog as a facilitator. In the CG, the same sessions will be conducted without the therapy dog. Assessment: UCLA Loneliness Scale, Goldberg Anxiety and Depression Scale, Emotional Well-Being Scale (e-CAP), Duke-UNC-11 Functional Social Support Questionnaire, and Satisfaction Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* People who are 65 years of age or older assigned to the Primary Health Care Center.
* With a diagnosis of "living alone" registered in the computerized clinical history.
* Present unwanted loneliness with a score higher than 3 on the Three-Item Loneliness Scale (TIL Scale). The TIL Scale consists of three questions: How often do you feel that you lack company?, How often do you feel excluded?, How often do you feel isolated? The response options consist of a three-level Likert scale: "almost never", "sometimes" and "often"; the results being from 3 to 9 points.
* Delivery of the information sheet and signature of the informed consent.

Exclusion Criteria:

* If in the initial interview they declared having allergy to dogs.
* Significant fear of dogs
* Meets research criteria for a diagnosis of dementia.
* Do not understand or speak Catalan or Spanish

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on UCLA (University of California at Los Angeles) scale at 9 weeks. | This scale was administered at baseline and at week 9
  The UCLA scale has proven to be a useful and sensitive instrument for measuring feelings of loneliness in the elderly. The scale consists of 10 questions scored between 1 and 4 points, allowing a minimum score of 10 and a maximum of 40.
  * Scores <20 may indicate a severe degree of loneliness.
  * Scores between 20-30 may indicate a moderate degree of loneliness.

SECONDARY OUTCOMES:
Change from baseline on Goldberg Anxiety and Depression Scale (GADS) at 9 weeks. | This scale was administered at baseline and at week 9
  The Goldberg anxiety and depression scale is an 18 item self-report symptom inventory with "yes" and "no" response options, with two subscales: one for anxiety (9 items) and one for depression (9 items). Higher scores mean a worse outcome.
Change from baseline on Emotional Well-Being Scale at 9 weeks. | This scale was administered at baseline and at week 9
  The questionnaire consists of seven items measured on a Likert scale, with five response options (1 = never and 5 = always) on how the individual has felt in the last two weeks; with a score range from 5 to 35, higher scores mean a better outcome.
Change from baseline on Duke-UNC-11 Functional Social Support Questionnaire at 9 weeks. | This scale was administered at baseline and at week 9
  The Duke-UNC-11 questionnaire assesses confidential social support (availability of people to communicate with) and affective social support (demonstrations of love, affection, and empathy). Likert scale with scores from 1 to 5. It consists of 11 items with a score range from 11 to 55 (a score <32 indicates low perceived social support)

OTHER OUTCOMES:
Satisfaction questionnaire at the end of the intervention at week 9 | This questionnaire was administered at week 9
  Satisfaction will be evaluated through a self-administered questionnaire to analyze the participants' satisfaction with the methodology, organization and resources, and the usefulness of the intervention. It will be scored on a 10-point Likert scale, from totally disagree to totally agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Atenció Primària Bordeta-Magraners, Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No